CLINICAL TRIAL: NCT06224777
Title: Comparison of Fluid Resuscitation in Pediatric Burn Patients Using Crystalloids and With Albumin on Day Two.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 260/RC/KEMU
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-09

CONDITIONS: Burns
Keywords: Albumin; Resuscitation; Pediatric Burns; Fluid creep; Shock; Crystalloids
MeSH Terms: conditions — Burns; Shock | interventions — Albumins; Solutions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albumin Group A (Experimental): 5% Albumin solution will be administered on day 2 @0.5ml/kg/%burn over 8 hours,in addition to required crystalloids.
  Interventions: Biological: 5% Albumin (human) Solution; Drug: Paeds solution
- Crystalloid Group B (Active Comparator): Routine Crystalloids will be administered according to weight of the patient.
  Interventions: Drug: Paeds solution

INTERVENTIONS:
Biological: 5% Albumin (human) Solution — Albumin is a biological product derived from human blood donors.
  Other Names: ALBURX® 5
  Arms: Albumin Group A
Drug: Paeds solution — Paeds solution contains dextrose 4.3%, and Sodium Chloride 0.18%
  Other Names: Revasol-Paeds IV Infusion

SUMMARY:
The goal of this comparative, interventional randomized controlled trial is to use albumin during resuscitation in pediatric burn patients on day 2, as it can reduce extravasation of fluids and decrease the overall fluid requirements, along with mortality and maintain circulation.

Participants will be divided into 2 groups. Albumin will be administered additionally in group A, while only crystalloids will be used for resuscitation in group B.

DETAILED DESCRIPTION:
The randomized controlled trial will be done at Department of Pediatric Surgery, Mayo Hospital Lahore from January 2022 to December 2022. Ninety patients (forty-five patients in each group) will be enrolled using a non probability convenient sampling technique. Patients will be randomly divided into 2 groups. Albumin solution will be administered in group A and in group B only routine crystalloids will be given. Basic demographic information will be noted. Effect modifiers (hemoglobin, Albumin level, weight and height) will be noted.

Group A: After first 24 hours, maintenance fluid, N/2+5%Dextrose solution will be started according to weight(100ml/kg/day for first 10kg, 50ml/kg/day for next 10kg and 20ml/kg/day for the remainder) and will be increased or decreased by 1/3 to maintain the urinary output to 1-1.5ml/kg/hour. 12, 75 5% Albumin solution will be administered @0.5ml/kg/%burn over initial 8 hours of day 2 and It's amount will be subtracted from the 24 hours fluid calculated earlier.

Group B: After first 24 hours, maintenance fluid, N/2+5%Dextrose solution will be started according to weight (100ml/kg/day for first 10kg, 50ml/kg/day for next 10kg and 20ml/kg/day for the remainder) and will be increased or decreased by 1/3 to maintain the urinary output to 1-1.5ml/kg/hour.

ELIGIBILITY:
Inclusion Criteria:

* 25-40%, less than 12 hours old, scald or flame burn patients
* Full thickness

Exclusion Criteria:

* Burns with inhalational injury.
* Patients hypersensitive to Albumin.
* Deranged renal or hepatic profile.
* Patients with known Cardiac or debilitating Congenital anomalies.
* Patients with known metabolic disease.
* Burns associated with trauma including fractures, head injuries, intra-abdominal bleed etc.
* Albumin level lower than 1.8g/dl at time of admission.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Resuscitation Volume | 24-48 hours
  Total volume of fluid required to maintain a urine output of 1-1.5ml/hour on the day 2 of admission.
Serum Albumin levels | 24-48 hours
  Albumin level in patient after day 2 of admission
Urine Output | 24-48 hours
  Amount of urine passed on day 2 of admission. Should be 1-2.5ml/kh/hr

SECONDARY OUTCOMES:
Requirement of inotropic support | 24-48 hours
  Patients in shock not responding to additional fluid administration, with reduced urine output requiring dopamine or dobutamine.
Mortality | First 5 days of admission
  Any death occuring within 5 days of admission

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Naumeri, MBBS,FCPS, Principal Investigator — King Edward Medical University
Locations (1):
- King Edward Medical University, Mayo Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romanowski KS, Palmieri TL. Pediatric burn resuscitation: past, present, and future. Burns Trauma. 2017 Sep 4;5:26. doi: 10.1186/s41038-017-0091-y. eCollection 2017. PMID 28879205
- [Background] O'Mara MS, Slater H, Goldfarb IW, Caushaj PF. A prospective, randomized evaluation of intra-abdominal pressures with crystalloid and colloid resuscitation in burn patients. J Trauma. 2005 May;58(5):1011-8. doi: 10.1097/01.ta.0000162732.39083.15. PMID 15920417
- [Background] Comish P, Walsh M, Castillo-Angeles M, Kuhlenschmidt K, Carlson D, Arnoldo B, Kubasiak J. Adoption of rescue colloid during burn resuscitation decreases fluid administered and restores end-organ perfusion. Burns. 2021 Dec;47(8):1844-1850. doi: 10.1016/j.burns.2021.02.005. Epub 2021 Feb 20. PMID 33658146
- See also: Rationale — https://pubmed.ncbi.nlm.nih.gov/28879205/